CLINICAL TRIAL: NCT05664113
Title: Feasibility, Safety, and Potential Efficacy of Fecal Microbiota Transplantation (FMT) for Gastrointestinal Dysfunction in Children Following Hematopoietic Cell Transplant (HCT).
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEWGUT; NCI-2024-02553 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gastro-Intestinal Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stratum A (Experimental): Diagnosed with GvHD
  Interventions: Drug: Fecal microbiota transplant (FMT)
- Stratum B (Experimental): GI Dysfunction
  Interventions: Drug: Fecal microbiota transplant (FMT)

INTERVENTIONS:
Drug: Fecal microbiota transplant (FMT) — FMT Lower Delivery Microbiota Preparation, Dose: 250 mL of Microbiota Preparation Material and Route of administration: colonoscopy FMT Upper Delivery Microbiota Preparation, Dose: 60 mL of Microbiota Preparation Material and Route of administration: Naso-enteral tube
  Other Names: FMT

SUMMARY:
The study participant is being asked to take part in this clinical trial, a type of research study, because the participant has Gastrointestinal (GI) symptoms following a Hematopoietic Cell Transplant (HCT).

Primary Objective

* To determine the safety and feasibility of FMT for treating a GvHD of the gut following HCT.
* To determine the safety and feasibility of FMT for treating HCT induced gut dysfunction.

Secondary Objectives

* To assess the potential efficacy of FMT for treating a GvHD of the gut following HCT.
* To assess the potential efficacy of FMT for treating HCT induced gut dysfunction.

DETAILED DESCRIPTION:
Participants will be eligible to receive an FMT on or after Day +30 post-HCT. FMT will be performed using FMP material obtained from OpenBiome. 60 mL of FMP will be administered via NJ tube and 250 mL via colonoscopy. A second FMT may be performed at least 14 days after the initial FMT in GI clinical symptoms have partially improved or have not changed. The second FMT will be administered using the same procedure as in the initial FMT

ELIGIBILITY:
Inclusion Criteria:

* Age < 22 years old.
* Received an allogeneic HCT greater than or equal to 30 days prior to enrollment
* Diagnosed with one of the following conditions:

  1. Steroid-resistant gut a GvHD (defined as GI symptoms that do not improve within 5 days after initial steroid therapy, >/= 1mg/kg of prednisolone) OR
  2. Steroid-dependent gut a GvHD (defined as the presence of a response to methylprednisolone 2 mg/kg/day but relapsing when an attempt was made to taper steroid treatment).

     OR
  3. Current or prolonged GI dysfunction following HCT, defined as having diarrhea or loose stools >/= 4 weeks with at least one of the following:

     1. Requiring NG or G-tube feeds
     2. Requiring TPN or IVF for more than 4 weeks
     3. Diagnosis of gastroparesis by GI specialist documented in the medical record
* Willing and able to provide informed assent/consent

Exclusion Criteria:

* Cytomegalovirus (CMV) or Epstein Barr Virus (EBV) IgG negative at the time of consent
* Female participant who is pregnant or nursing
* History of previous FMT
* Intra-abdominal surgery within 4 weeks of enrollment
* At increased risk for peritonitis: presence of intra-abdominal devices (G-or GJ-tubes are acceptable), receiving peritoneal dialysis, or ascites
* Concurrent abdominal radiation therapy
* Any acute or chronic illness/condition as well as medication that in the opinion of the investigator puts the subject at greater risk from FMT or may confound the study results.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a serious adverse event occurring within 30 days following FMT | 30 Days
  Serious adverse events will be a primary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction
Proportion of participants with a non-serious adverse event occurring within 30 days following FMT | 30 Days
  Non-serious adverse events will be a primary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction
Proportion of patients expressing interest who meet eligibility | 2 years
  Participant eligibility will be a primary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction
Proportion of patients recruited in the eligible population | 2 years
  Participant recruitment will be a primary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction
Proportion of participants that drop up post-enrollment | 3 years
  Participant retention will be a primary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction
Proportion of participants providing all protocol required stool samples | 3 years
  Stool specimens will be a primary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction

SECONDARY OUTCOMES:
Proportion of participants with a complete response or a partial response | 180 days
  Complete response or partial response will be a secondary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction
Percentage of participants who reduce or discontinue steroids at the end of the study | 1 year
  Reduction in dose of steroids will be a secondary outcome measure for the following groups:
  * FMT for treating a GvHD of the gut following HCT
  * FMT for treating HCT induced gut dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Maron, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols